CLINICAL TRIAL: NCT03425747
Title: CALCIUM CITRATE vs CALCIUM CARBONATE FOR THE MANAGEMENT OF CHRONIC HYPOPARATHYROIDISM
Brief Title: Efficacy of Calcium Citrate Versus Calcium Carbonate for the Management of Chronic Hypoparathyroidism
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Campus Bio-Medico University (Other)
Responsible Party: Principal Investigator, Andrea Palermo, Principal Investigator, Campus Bio-Medico University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Ca Citrate VS Ca Carbonate
Record Dates: First submitted 2018-01-27; First posted 2018-02-08 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Chronic Hypoparathyroidism
Keywords: calcium carbonate; calcium citrate; quality of life; hypoparathyroidism; hypocalcemia; calicum oxalate saturation; kydney stone
MeSH Terms: conditions — Hypoparathyroidism; Hypocalcemia | interventions — Calcium Carbonate; Calcium Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calcium Carbonate (Active Comparator): Calcium Carbonate
  Interventions: Drug: Calcium Carbonate; Drug: Calcium Citrate
- calcium Citrate (Active Comparator): Calcium Citrate
  Interventions: Drug: Calcium Carbonate; Drug: Calcium Citrate

INTERVENTIONS:
Drug: Calcium Carbonate — subjects will be assigned to a calcium supplement (Carbonate or Citrate) at the same total amount of elemental calcium that they had taken before the study enrolment.
Drug: Calcium Citrate — subjects will be assigned to a calcium supplement (Carbonate or Citrate) at the same total amount of elemental calcium that they had taken before the study enrolment.

SUMMARY:
Hypoparathyroidism is an endocrinopathy characterized by a deficient secretion or action of PTH associated with low calcium level. According to the European guideline (2015), standard treatment includes oral calcium salts and active vitamin D metabolites to relieve symptoms of hypocalcaemia, maintain serum calcium levels in the low normal range and improve the patient's QoL Calcium carbonate is most often used and less expensive than other calcium preparations and contains the highest concentration of elemental calcium per gram (42%). It requires gastric hydrochloric acid to form carbonic acid (H2CO3) that immediately decomposes into water (H2O) and carbon dioxide (CO2). CO2 is responsible for its side effects such as flatulence, constipation and general gastrointestinal disorders. Therefore, in some patients it is better to find an alternative to calcium carbonate. Calcium citrate should be recommended to patients with achlorhydria or on treatment with proton pump inhibitors (PPI) as well as to patients who preferred to take supplements outside mealtimes. furthermore, patients with hypoparathyroidism have an increased risk of kidney stones. Kidney stones are formed by calcium salts, among which the most frequent ones are calcium-oxalate (70-80%), followed by calcium-phosphate and uric acid. Citrate salts are widely used in the treatmentof nephrolithiasis, since have shown an inhibitory effect on kidney stone formation. Up to now, there are no studies aimed to investigate the efficacy of calcium citrate in the management of subjects with chronic hypoparathyroidism. In particular, we will investigate if calcium citrate compared to calcium carbonate does not affect the risk of renal stones, if it is able to maintain normal calcium levels and, if it has an impact on QOL, in subjects with chronic hypoparathyroidism.

DETAILED DESCRIPTION:
BACKGROUND Hypoparathyroidism is an endocrinopathy characterized by a deficient secretion or action of PTH associated with low calcium level. It can be primary (inadequate PTH activity), or secondary (peripheral resistance to PTH).

The most common cause of chronic Hypoparathyroidism is the postsurgical one: it is usually secondary to previous thyroid surgery but may also occur following parathyroidectomy or other cervical surgical procedures. Transient Hypoparathyroidism occurs in 30-60% of patients undergoing total or subtotal thyroidectomy. About 60-70% of cases of postoperative hypocalcaemia resolve within 4-6 weeks after surgery. About 15-25% of patients will develop chronic Hypoparathyroidism. The risk of chronic Hypoparathyroidism is closely related to the number of parathyroid glands remaining in situ at operation.

Hypocalcemia is defined as serum calcium level (albumin adjusted total calcium or ionized calcium) below the lower limit of the reference range (target range).

In literature there are not data that suggest which is the best serum calcium level to maintain during treatment, but the aim is to maintain serum calcium level in the lower part or slightly below the lower limit of the reference range (adjusted serum calcium level <2.1-2.3 or S-Ca2+ between 1.05-1.15mmol/L), serum phosphate levels within the reference range, serum calcium-phosphate product below 4.4 mmol2/l2 (55 mg2/dl2), 24-hurinary calcium excretion <7.5 mmol/2h (300 mg/24h) in men, <6.25 mmol/24h (250 mg/24h) in women, or <0.1 mmol/kg per 24 h (4 mg/kg per 24h) in both sexes.

In addition to hypocalcemia, patients affected by chronic hypoparathyroidism have a higher risk of renal implications such as urolithiasis and renal impairment because lack of PTH reduces calcium absorption and phosphate excretion causing hypercalciuria and hyperphosphatemia.

Moreover, many patients with hypoparathyroidism complain of reduced quality of life (QOL) in ways that are difficult to quantify but that are nevertheless of concern. Biochemical control with standard therapy is rarely accompanied by improved functioning or sense of well-being. Complaints of cognitive dysfunction are common, with the term brain fog typically described by patients. In support of these issues, large cohort studies from Denmark have shown increased risk of hospitalization for depression and affective disorders, renal impairment and infections, whereas the risk for cancer and overall mortality was not increased.

According to the European guideline (2015), standard treatment includes oral calcium salts and active vitamin D metabolites to relieve symptoms of hypocalcaemia, maintain serum calcium levels in the low normal range and improve the patient's QoL An adequate daily intake of calcium from diet and supplements is advisable. Different calcium salts are available as supplements because elemental calcium is highly reactive so it has to be combined with other substances. These preparations differ in the concentration of elemental calcium per gram.

Calcium carbonate is most often used and less expensive than other calcium preparations and contains the highest concentration of elemental calcium per gram (42%). It requires gastric hydrochloric acid to form carbonic acid (H2CO3) that immediately decomposes into water (H2O) and carbon dioxide (CO2). CO2 is responsible for its side effects such as flatulence, constipation and general gastrointestinal disorders. Therefore, in some patients it is better to find an alternative to calcium carbonate. Calcium citrate, for example, should be recommended to patients with achlorhydria or on treatment with proton pump inhibitors (PPI) as well as to patients who preferred to take supplements outside mealtimes.

Previous studies showed that calcium citrate, in comparison to calcium carbonate, causes greater increment in serum calcium concentration and urinary calcium excretion in parallel with greater suppression of serum PTH, after Roux-en-Y Gastric bypass and this datum suggests both the pharmacokinetic and pharmacodynamic superiority of calcium citrate.

Calcium citrate is also better adsorbed than calcium carbonate after panproctocolectomy, so in a condition of a general enteric malabsorption.

Up to now, there are no studies aimed to investigate the efficacy of calcium citrate in the management of subjects with chronic hypoparathyroidism. In particular, the investigators will test the efficacy of calcium citrate in maintaining normal calcium level compared to carbonate calcium in subjects with chronic hypoparathyroidism. Moreover, the investigators will evaluate the impact of calcium citrate on QOL in this kind of patients compared to the gold standard therapy (carbonate calcium).

MATERIALS AND METHODS Each subject will participate in two phases of the study and each phase will last one month. Once every 2 weeks blood and a morning urine sample will be drawn. For all the study period, participants will be instructed to maintain a predetermined dietary calcium intake (800 mg/day) with sodium (100 mEq/day) restrictions. All subjects will complete a questionnaire on quality of life at 0, +2, +4 week, during both phases. The investigators will use the Rand 36-Item Short Form Health Survey (version 1.0) to evaluate the QOL.

Phase 1: According to a block randomization scheme, subjects will be assigned to a calcium supplement (Drug A or Drug B) at the same total amount of elemental calcium that they had taken before the study enrollment. The dose of Vitamin D will be equal to the daily dose taken prior to the study, and will not be changed during the study period.

Phase 2: subjects will be shift to the opposite Drug (from drug A to drug B or from drug B to drug A) at the same total amount of elemental calcium that they had taken during the last week of the phase 1.

SAMPLE SIZE CALCULATION

1. Based on the assumption that the within-patient standard deviation of the calcium oxalate saturation is 0.5, to demonstrate that calcium citrate does not affect the calcium oxalate saturation, a total of 24 patients need to be enrolled in this study. This sample size will allow to detect a difference of 0.43 points at a two-sided 5% significance level with a probability of type II error of 20%.
2. to demonstrate that calcium citrate is as effective as calcium carbonate in maintaining serum Ca within the acceptable clinical range. To this end, we will study a sample of 21 people already treated with calcium and vitamin D supplementation. Our hypothesis is that at the end of the study period, the mean Ca concentration will not be different from the ideal value (9 mg/dl), accepting a 10% variation as the equivalence limit (i.e., accepting as equivalent values between 8.1 and 9.9 mg/dl). Under these assumptions, we would need 11 patients to show equivalence between the two treatments, with a alpha error probability of 5% and a beta error probability of 10%20. With the available sample size, we will be able to establish equivalence with an equivalence limit of 0.7 (i.e., values between 8.3 and 9.7 mg/dl).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of postsurgical chronic hypoparathyroidism by at least 6 months
* No change of treatment over the last 3 months prior to enrollment.
* Values of serum calcium and phosphorus stable over the last three months prior to enrollment
* Absence of symptoms from hypocalcaemia in the 3 months prior to enrollment
* A requirement for active vitamin D (calcitriol ≥0.25 mcg daily) and oral calcium (≥1000 mg daily) treatment.

Exclusion Criteria:

* liver failure
* renal failure (gfr <30 ml/min)
* hypercalcemia
* hyperthyroidism
* parathyroid disorders
* use of the following drugs within 3 months of the study: diuretics, bisphosphonates, calcitonin, corticosteroids, anabolic steroids, anticonvulsants, H2 receptor antagonists or proton pump inhibitor
* heavy smokers (>10 cigarettes/day)
* abusing alcohol (>70 ml/day)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Change in serum calcium level | 0, 1 and 2 months
  albumin-adjusted calcium levels
Change in calcium oxalate saturation | 0, 1 and 2 months
  24-h urinary calcium oxalate saturation

SECONDARY OUTCOMES:
Change in Quality of life and fatigue | 0,1,2 months
  PCS and MCS (by SF-36 survey) and fatigue score

CONTACTS AND LOCATIONS:
Locations (1):
- Campus Bio-Medico University, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cusano NE, Rubin MR, Bilezikian JP. Parathyroid hormone therapy for hypoparathyroidism. Best Pract Res Clin Endocrinol Metab. 2015 Jan;29(1):47-55. doi: 10.1016/j.beem.2014.09.001. Epub 2014 Sep 10. PMID 25617172
- [Background] Shoback D. Clinical practice. Hypoparathyroidism. N Engl J Med. 2008 Jul 24;359(4):391-403. doi: 10.1056/NEJMcp0803050. No abstract available. PMID 18650515
- [Background] Bollerslev J, Rejnmark L, Marcocci C, Shoback DM, Sitges-Serra A, van Biesen W, Dekkers OM; European Society of Endocrinology. European Society of Endocrinology Clinical Guideline: Treatment of chronic hypoparathyroidism in adults. Eur J Endocrinol. 2015 Aug;173(2):G1-20. doi: 10.1530/EJE-15-0628. PMID 26160136
- [Background] Cusano NE, Rubin MR, McMahon DJ, Irani D, Tulley A, Sliney J Jr, Bilezikian JP. The effect of PTH(1-84) on quality of life in hypoparathyroidism. J Clin Endocrinol Metab. 2013 Jun;98(6):2356-61. doi: 10.1210/jc.2013-1239. Epub 2013 Apr 17. PMID 23596139
- [Background] Arlt W, Fremerey C, Callies F, Reincke M, Schneider P, Timmermann W, Allolio B. Well-being, mood and calcium homeostasis in patients with hypoparathyroidism receiving standard treatment with calcium and vitamin D. Eur J Endocrinol. 2002 Feb;146(2):215-22. doi: 10.1530/eje.0.1460215. PMID 11834431
- [Background] Bilezikian JP, Khan A, Potts JT Jr, Brandi ML, Clarke BL, Shoback D, Juppner H, D'Amour P, Fox J, Rejnmark L, Mosekilde L, Rubin MR, Dempster D, Gafni R, Collins MT, Sliney J, Sanders J. Hypoparathyroidism in the adult: epidemiology, diagnosis, pathophysiology, target-organ involvement, treatment, and challenges for future research. J Bone Miner Res. 2011 Oct;26(10):2317-37. doi: 10.1002/jbmr.483. PMID 21812031
- [Background] Harvey JA, Zobitz MM, Pak CY. Dose dependency of calcium absorption: a comparison of calcium carbonate and calcium citrate. J Bone Miner Res. 1988 Jun;3(3):253-8. doi: 10.1002/jbmr.5650030303. PMID 3213620
- [Background] Straub DA. Calcium supplementation in clinical practice: a review of forms, doses, and indications. Nutr Clin Pract. 2007 Jun;22(3):286-96. doi: 10.1177/0115426507022003286. PMID 17507729
- [Background] Tondapu P, Provost D, Adams-Huet B, Sims T, Chang C, Sakhaee K. Comparison of the absorption of calcium carbonate and calcium citrate after Roux-en-Y gastric bypass. Obes Surg. 2009 Sep;19(9):1256-61. doi: 10.1007/s11695-009-9850-6. Epub 2009 May 13. PMID 19437082
- [Background] Santonati A, Palermo A, Maddaloni E, Bosco D, Spada A, Grimaldi F, Raggiunti B, Volpe R, Manfrini S, Vescini F; Hypoparathyroidism AME Group. PTH(1-34) for Surgical Hypoparathyroidism: A Prospective, Open-Label Investigation of Efficacy and Quality of Life. J Clin Endocrinol Metab. 2015 Sep;100(9):3590-7. doi: 10.1210/jc.2015-1855. Epub 2015 Jul 21. PMID 26196949
- [Background] Cusano NE, Rubin MR, McMahon DJ, Irani D, Anderson L, Levy E, Bilezikian JP. PTH(1-84) is associated with improved quality of life in hypoparathyroidism through 5 years of therapy. J Clin Endocrinol Metab. 2014 Oct;99(10):3694-9. doi: 10.1210/jc.2014-2267. Epub 2014 Jun 30. PMID 24978675